CLINICAL TRIAL: NCT02419807
Title: Comparison of Use of Indocyanine Green and 99mTc-labeled Radiotracer for Axillary Lymphatic Mapping in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mitaka USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE10114
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Stage I Breast Cancer; Stage II Breast Cancer
Keywords: Near Infrared Fluorescence Imaging; Indocyanine Green; axillary lymph node mapping; Mastectomy, Segmental; Sentinel Lymph Node Biopsy; Lumpectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (indocyanine green, 99mTc-labeled radiotracer) (Experimental): Participants receive technetium Tc-99m sulfur colloid injection and undergo lymphoscintigraphy according to clinical practice. Prior to surgery, participants also receive indocyanine green solution subdermally close to the tumor or into subareolar region of the breast skin. Participants then undergo Axillary Lymph Node Biopsy and surgery.
  Interventions: Drug: Indocyanine Green Solution; Radiation: Technetium Tc-99m Sulfur Colloid; Procedure: Lymphoscintigraphy; Procedure: Axillary Lymph Node Biopsy

INTERVENTIONS:
Drug: Indocyanine Green Solution — Given subdermally
  Other Names: IC-GREEN; ICG solution
Radiation: Technetium Tc-99m Sulfur Colloid — Given via injection
  Other Names: Tc 99m Sulfur Colloid; Tc-99m SC; Technetium Tc 99m Sulfur Colloid
Procedure: Lymphoscintigraphy — This is a method used to check the lymph system for disease. A radioactive substance that flows through the lymph ducts and can be taken up by lymph nodes is injected into the body. A scanner or probe is used to follow the movement of this substance on a computer screen. Lymphoscintigraphy is used to find the sentinel lymph node (the first node to receive lymph from a tumor), which may be removed and checked for tumor cells. Lymphoscintigraphy is also used to diagnose certain diseases or conditions, such as lymphoma or lymphedema.
  Other Names: Undergo lymphoscintigraphy
Procedure: Axillary Lymph Node Biopsy — Undergo biopsy
  Other Names: Axillary Node Biopsy; axillary sentinel lymph node biopsy

SUMMARY:
This clinical trial will enroll up to 130 adult women with a confirmed diagnosis of clinical stage 1 or 2 breast cancer who are undergoing breast cancer surgery with lumpectomy or mastectomy and planned axillary sentinel node biopsy procedure. Participants will undergo lymphatic mapping with technetium Tc-99m (99mTc) sulfur colloid in accordance with routine clinical practice. Injections of 99mTc sulfur colloid will take place the afternoon prior to planned next morning surgery or on the morning of surgery. Participants will undergo lymphoscintigraphy in accordance with standard clinical practice.

Immediately prior to operation, after the induction of anesthesia in the operating room, up to 1cc of 0.5% indocyanine green (ICG) solution will be injected subdermally close to the tumor or into the subareolar region after disinfection of the breast skin. ICG movement will be facilitated by manual massage and monitored with fluorescence imaging. ICG fluorescence will be elicited and detected by Photodynamic Eye (PDE) camera. The lymphatic drainage, made evident by the fluorescent dye, will be monitored in real time on a monitor. The fluorescence will be followed towards the armpit region (axilla) and time for the fluorescence to reach the axilla will be recorded. Following standard practice, an incision will be made in the armpit region. Fluorescent lymph nodes (ICG positive) will be localized and removed and analyzed by a pathologist. Node removal will continue until no residual fluorescence is visible in the axilla. Removed nodes will be tested for radioactivity using a standard gamma-detecting probe and the counts per minute will be recorded. Finally, the armpit region will be inspected with the gamma probe to determine if there are any residual radioactive nodes. Residual sentinel nodes (the first node to receive lymph from a tumor) will be removed. For the purposes of this study, the sentinel status of a node will be defined as being flagged as sentinel by either one or both of the ICG or 99mTc methods. The goal of the project is to confirm that axillary lymphatic mapping with ICG leads to similar nodes being labeled as sentinel as lymphatic mapping with 99mTc-labeled radiotracer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm that axillary lymphatic mapping with indocyanine green solution (ICG) solution leads to a similar number of nodes being labeled as sentinel as lymphatic mapping with 99mTc-labeled (technetium Tc-99m sulfur colloid) radiotracer.

OUTLINE:

Participants receive technetium Tc-99m sulfur colloid injection and undergo lymphoscintigraphy according to clinical practice. Prior to surgery, participants also receive indocyanine green solution subdermally close to the tumor or into subareolar region of the breast skin. Participants then undergo axillary sentinel node biopsy and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a confirmed diagnosis of clinical stage 1 or 2 breast cancer
* Participants who are undergoing breast cancer surgery with lumpectomy or mastectomy
* Participants with planned axillary sentinel node biopsy procedure

Exclusion Criteria:

* Participants with cancer > 3 cm
* Participants with clinically positive nodes
* Participants with prior surgery for breast cancer in the index breast
* Participants who have had bilateral breast surgeries
* Thyroid dysfunction
* Hypersensitivity to iodine
* Hepatic insufficiency
* Renal insufficiency

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Grobmyer, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Instititute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Indocyanine Green, 99mTc-labeled Radiotracer)
Started | 102
Completed | 92
Not Completed | 10
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Population: Participants who enrolled on study
Arm/Group | Diagnostic (Indocyanine Green, 99mTc-labeled Radiotracer)
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 90
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 102
Tc-positive and ICG-positive sentinel nodes (SNs) [Number; unit: sentinel nodes] | 191
Tc-positive and ICG-negative sentinel nodes (SNs) [Number; unit: sentinel nodes] | 11
Tc-negative and ICG-positive SNs [Number; unit: sentinel nodes] | 33
Total sentinel lymph nodes (SLNs) [Number; unit: sentinel nodes] | 235

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Sentinel Lymph Nodes (SLNs) Flagged by the Two Methods
Description: Let A be the number of Tc-positive and ICG-positive sentinel nodes (SNs) detected, B be the number of Tc-positive and ICG-negative SNs detected, and C be the number of Tc-negative and ICG-positive SNs detected. The total number (N) of SNs detected is therefore N = (A + B + C); the proportion of SNs detected by the Tc method (PTc) is (A + B)/N; and the proportion of SNs detected by the ICG method (PICG) is (A + C)/N. Differences in the proportions of SLNs flagged will be compared using a two-sided 95% confidence interval.
Time Frame: Baseline
Population: Participants who completed study
Measure: Number; unit: proportion of nodes
Arm/Group | Diagnostic (Indocyanine Green, 99mTc-labeled Radiotracer)
Number analyzed (Participants) | 92
proportion of nodes
  Proportion of SNs (PTc) detected by Tc method | 0.86
  Proportion of SNs (PICG) detected by ICG method | 0.95
Statistical Analysis 1: Comparison: Diagnostic (Indocyanine Green, 99mTc-labeled Radiotracer); Test type: Equivalence — Equivalence is defined as the difference in the proportions of nodes flagged between the Tc and ICG methods falling within an interval (-δ, +δ), where δ is taken to be 5%; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.036 to 0.151]

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events for 30 days following their surgical operation
Arm/Group | Diagnostic (Indocyanine Green, 99mTc-labeled Radiotracer)
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT02419807/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT02419807/ICF_001.pdf